CLINICAL TRIAL: NCT03140930
Title: The Effect of Duodenal, Ileal or Combined Infusion of Tastants on Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Tim Klaassen, MD, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NL59530.068.16
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Duodenal tastants, ileal placebo (Experimental): Duodenal infusion of combination of tastants (sweet, bitter and umami), ileal infusion of placebo (tap water)
  Interventions: Dietary Supplement: Tastants duodenal; Dietary Supplement: Placebo ileal
- Duodenal placebo, ileal tastants (Experimental): Duodenal infusion of placebo (tap water), ileal infusion of combination of tastants (sweet, bitter and umami)
  Interventions: Dietary Supplement: Tastants ileal; Dietary Supplement: Placebo duodenal
- Duodenal tastants, ileal tastants (Experimental): Duodenal infusion of combination of tastants (sweet, bitter and umami), ileal infusion of combination of tastants (sweet, bitter and umami)
  Interventions: Dietary Supplement: Tastants duodenal; Dietary Supplement: Tastants ileal
- Duodenal placebo, ileal placebo (Placebo Comparator): Duodenal infusion of placebo (tap water), ileal infusion of placebo (tap water)
  Interventions: Dietary Supplement: Placebo duodenal; Dietary Supplement: Placebo ileal

INTERVENTIONS:
Dietary Supplement: Tastants duodenal — Duodenal infusion of combination of tastants (sweet, bitter and umami)
  Arms: Duodenal tastants, ileal placebo; Duodenal tastants, ileal tastants
Dietary Supplement: Tastants ileal — Ileal infusion of combination of tastants (sweet, bitter and umami)
  Arms: Duodenal placebo, ileal tastants; Duodenal tastants, ileal tastants
Dietary Supplement: Placebo duodenal — Duodenal infusion of placebo (tap water)
  Arms: Duodenal placebo, ileal placebo; Duodenal placebo, ileal tastants
Dietary Supplement: Placebo ileal — Ileal infusion of placebo (tap water)
  Arms: Duodenal placebo, ileal placebo; Duodenal tastants, ileal placebo

SUMMARY:
Rationale: The appearance of tastants in the small intestine can result in the activation of a negative feedback mechanism from different parts of the intestine to the stomach, the small intestine and to the central nervous system. These processes inhibit food processing, appetite sensations and food intake, and furthermore they increase feelings of satiety and satiation. The effects of intraduodenal and/or intraileal infusion of a combination of tastants (sweet (rebaudioside A), bitter (quinine) en umami (monosodium glutamate(MSG))) and placebo on ad libitum food intake, satiation and gastrointestinal symptoms will be investigated.

Objective: To investigate the effect of intraduodenal, intraileal and combined infusion of a combination of tastants versus infusion of placebo on food intake.

Secondary objectives:

1. To compare the effect of intraduodenal versus intraileal versus combined intraduodenal and intraileal delivery of a combination of tastants on satiation.
2. To assess the effect of intraduodenal and/or intraileal delivery of a combination of tastants on gastrointestinal symptoms/complaints.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous examination, no gastrointestinal complaints can be defined.
* Age between 18 and 65 years. This study will include healthy adult subjects (male and female). Women must be taking contraceptives.
* BMI between 18 and 25 kg/m2)
* Weight stable over at least the last 6 months

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided by the principal investigator.
* Use of medication, including vitamin supplementation, except oral contraceptives, within 14 days prior to testing
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principle investigator)
* Dieting (medically prescribed, vegetarian, diabetic, microbiological, biological dynamic)
* Pregnancy, lactation
* Excessive alcohol consumption (>20 alcoholic consumptions per week)
* Smoking
* Weight <60kg
* Non-tasters of sweet, bitter or umami
* Evidence of MSG-hypersensitivity or Chinese restaurant syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Ad libitum meal intake | 5 weeks
  Difference in ad libitum meal intake (as measured during ad libitum pasta meal) at end of the test day.

SECONDARY OUTCOMES:
Satiation | 5 weeks
  Difference in satiation (as measured by VAS) per time point.
GI-symptoms | 5 weeks
  Difference in gastro-intestinal symptoms (as measured by VAS) per time point.

CONTACTS AND LOCATIONS:
Overall Officials: Ad AM Masclee, Prof., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No